CLINICAL TRIAL: NCT06667869
Title: Sistema de monitorización multiparámetros Para sedación de Pacientes críticos en UCI (ROMANTIC: multipaRameter mOnitoring systeM for sedAtion iNThe ICu)
Brief Title: multipaRameter mOnitoring systeM for sedAtion iNThe ICu
Acronym: ROMANTIC
Status: Recruiting | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Agencia Nacional de Investigacion y Desarrollo, ANID (Unknown)
Responsible Party: Sponsor
Other Study IDs: 230926014; FONDEF ID24I10057 (Other Grant/Funding Number: Agencia Nacional de Investigación y Desarrollo)
Record Dates: First submitted 2024-09-30; First posted 2024-10-31 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-02

CONDITIONS: Sedation Complication
Keywords: Intensive Care Unit; Machine Learning; Delirium; Mechanical ventilation; Monitoring
MeSH Terms: conditions — Delirium | interventions — Hypnotics and Sedatives; Respiration, Artificial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Biospecimen Retention: Samples Without DNA — Blood samples for sedatives quantification
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Hospital Clínico Red de Salud UC-Christus: Adult patients admitted to intensive care units at Hospital Clinico Red de Salud UC-Christus who require sedation and mechanical ventilation for more than 24 hours.
  Interventions: Drug: Sedative
- Hospital Dr. Sotero del Rio: Adult patients admitted to intensive care units at Hospital Dr. Sotero del Rio who require sedation and mechanical ventilation for more than 24 hours.
  Interventions: Drug: Sedative

INTERVENTIONS:
Drug: Sedative — Patients admitted to intensive care units who require sedation and mechanical ventilation for more than 24 hours.
  Other Names: Mechanical ventilation

SUMMARY:
The administration of sedation in Intensive Care Units (ICU) is a vital and complex task, essential for the well-being of critically ill patients. Proper dosing is crucial, as both under-dosing and overdosing have adverse consequences for patients, including risks such as accidental extubation, ventilator disconnections, delirium, prolonged ventilation, ICU stays, and even increased mortality.

Monitoring sedation levels is essential to maintain a balance in sedative administration. Clinical scales (RASS/SAS) are currently used as the reference method, but they have limitations. These scales may be inadequate when the patient is unresponsive or when neuromuscular blockers are used. An alternative is electroencephalography (EEG)-based monitors, though they also have limitations in accurately representing the level of hypnosis.

The proposal is to develop an advanced multiparameter system called ROMANTIC, which utilizes machine learning algorithms to monitor sedation status continuously. The aim is for this system to surpass current techniques and provide a more accurate determination of sedation levels. ROMANTIC would incorporate a variety of variables, demographic, pharmacological, hemodynamic, respiratory, and EEG data, to predict sedation status in three categories: under-dosing, appropriate dosing, and overdosing.

With ROMANTIC, clinical staff (users) are expected to be able to determine sedation levels more quickly and accurately, reducing patients' wake-up times and possibly decreasing the incidence of delirium. In the long term, this could result in fewer ICU bed days, less time on mechanical ventilation, cost savings, and reduced complications.

At the end of the project, the goal is to have a prototype model or software that allows non-specialized staff (users) to quickly determine sedation levels in the ICU. This machine learning-based model targets hospitals with ICUs and mechanical ventilation to offer more efficient and cost-effective clinical care. ROMANTIC seeks to innovate in sedation monitoring, providing a more advanced and precise tool for the care of critically ill patients (beneficiaries) in the ICU.

DETAILED DESCRIPTION:
The project is characterized by incorporating multiple clinical, demographic, and pharmacological variables, along with prediction methods based on machine learning, to classify the level of sedation of critically ill patients into three broad categories: underdosage, appropriate dosage, and overdosage. The investigators will compare the performance of this approach against the current gold standard, which is the use of validated clinical sedation scales (RASS/SAS).

The design of this project is divided into two phases. The first phase involves a prospective observational cohort study where demographic, vital signs, ventilatory, pharmacological, and EEG variables will be collected from ICU patients. The second phase involves using the data obtained to create a multiparameter model with machine learning tools that informs ICU staff about the depth of sedation or the degree of hypnosis of each patient. Data will be collected from two national intensive care units: Hospital Clinico Red UC-CHRISTUS (associated entity) and Dr. Sótero del Río Hospital (associated entity). A technical team specialized in data collection and analysis, clinical research, and algorithm development from Pontificia Universidad Católica de Chile (beneficiary entity) will use this information to create a retrospective classifier that categorizes patients into one of three groups: underdosed, appropriately dosed, and overdosed.

Upon admission, comprehensive patient data will be collected, including age, sex, cause of connection to mechanical ventilation, comorbidities, and educational level. The researchers will also record the drugs and doses used for sedation, neuromuscular relaxants, and vasopressor drugs. Sedation will be administered with Fentanyl plus Propofol or Midazolam, according to usual clinical practices at both participating centers. Data from the RASS and SAS clinical sedation rating scales will be collected every hour during two time windows, providing a detailed picture of the patient's sedation levels.

There will be two or three data recording windows per patient. Time zero will be when the patient is intubated and connected to mechanical ventilation. The first collection window will be between 18 to 60 hours after intubation, for a period of 6 hours during business hours, aiming to obtain a record of data once the chosen sedation strategy is established and has presumably stable blood levels of drugs. The second window will start once the patient's sedation is suspended and will last for at least 6 hours or until the patient awakens, defined as SAS 4 and RASS 0, with eyes open to verbal command or if the patient presents agitation and/or delirium according to CAM-ICU. The suspension time will be recorded, along with the day and time all sedatives are stopped in the continuous infusion pump. If for any reason it is necessary to sedate the patient again, a third window similar to the second will be performed.

Demographic (age, previous educational level, SOFA, Charlson, APACHE II), hemodynamic (systolic and diastolic blood pressure, heart rate, electrocardiography), ventilatory (oxygen saturation, respiratory rate, ventilatory mode, PEEP, tidal volume, plateau pressure, peak pressure), electroencephalographic (EEG signal in time domain), pain (hourly behavioral pain scale), neuromuscular blockade (hourly TOF), and pharmacological (total mass of sedative drugs used at the time of suspending infusions and plasma samples of sedative drug concentration at the beginning of both windows) data will be collected. Once patients wake up, the onset of delirium will be assessed with the CAM-ICU tool twice a day (AM/PM) by appropriately trained nursing staff.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to adult critical care units
* Individuals over 18 years old
* Requiring sedation for more than 24 hours
* Patients needing mechanical ventilation for more than 24 hours

Exclusion Criteria:

* Patients with neurological pathology as the cause of mechanical ventilation (including recovered cardiocirculatory arrest, fulminant liver failure, and neurocritical conditions, except subdural hematomas or subarachnoid hemorrhages).
* Pregnancy
* Presence of psychiatric or intellectual disability prior to hospitalization
* Drug dependency
* History of chronic liver damage with hepatic encephalopathy
* Second period of mechanical ventilation during hospitalization
* Early limitation of therapeutic effort
* Patients under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to intensive care units requiring sedation and mechanical ventilation for more than 24 hours.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Time to extubation | From the start of last window up to extubation (assessed up to 72 hours)
  Time elapsed from the stop of sedative drugs to extubation (assessed up to 72 hours)

SECONDARY OUTCOMES:
Length of Intensive Care Unit stay | During intensive care unit hospitalization (assessed up to 100 days)
  Time (assessed up to 100 days) elapsed from admission to discharge from intensive care unit
Length of mechanical ventilation | During intensive care unit hospitalization (assessed up to 100 days)
  Time (assessed up to 100 days) elapsed from intubation to extubation
Intensive Care Unit Delirium incidence | From extubation to discharge from Intensive Care Unit, CAM-ICU assessed twice daily (AM/PM) for the first 5 post extubation days
  Positive Confusion Assessment Method for the Intensive Care Unit (CAM-ICU)
Serum concentration of sedative drugs | At baseline of all data extraction windows (assessed at the first hour of the respective window)
  Quantification of serum concentration of sedative drugs (Midazolam, Propofol, Fentanyl)

CONTACTS AND LOCATIONS:
Overall Officials: Juan C. Pedemonte, M.D., Study Director — Pontificia Universidad Catolica de Chile
Locations (2):
- Chile (2):
  - Hospital Dr. Sotero del Rio, Santiago, Metropolitana de Santiago
  - Hospital Clínico Pontificia Universidad Católica de Chile, Santiago, Santiago Metropolitan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Erstad BL, Puntillo K, Gilbert HC, Grap MJ, Li D, Medina J, Mularski RA, Pasero C, Varkey B, Sessler CN. Pain management principles in the critically ill. Chest. 2009 Apr;135(4):1075-1086. doi: 10.1378/chest.08-2264. PMID 19349403
- [Background] Rotondi AJ, Chelluri L, Sirio C, Mendelsohn A, Schulz R, Belle S, Im K, Donahoe M, Pinsky MR. Patients' recollections of stressful experiences while receiving prolonged mechanical ventilation in an intensive care unit. Crit Care Med. 2002 Apr;30(4):746-52. doi: 10.1097/00003246-200204000-00004. PMID 11940739
- [Background] Jackson DL, Proudfoot CW, Cann KF, Walsh T. A systematic review of the impact of sedation practice in the ICU on resource use, costs and patient safety. Crit Care. 2010;14(2):R59. doi: 10.1186/cc8956. Epub 2010 Apr 9. PMID 20380720
- [Background] Reade MC, Finfer S. Sedation and delirium in the intensive care unit. N Engl J Med. 2014 Jan 30;370(5):444-54. doi: 10.1056/NEJMra1208705. No abstract available. PMID 24476433
- [Background] Devlin JW, Skrobik Y, Gelinas C, Needham DM, Slooter AJC, Pandharipande PP, Watson PL, Weinhouse GL, Nunnally ME, Rochwerg B, Balas MC, van den Boogaard M, Bosma KJ, Brummel NE, Chanques G, Denehy L, Drouot X, Fraser GL, Harris JE, Joffe AM, Kho ME, Kress JP, Lanphere JA, McKinley S, Neufeld KJ, Pisani MA, Payen JF, Pun BT, Puntillo KA, Riker RR, Robinson BRH, Shehabi Y, Szumita PM, Winkelman C, Centofanti JE, Price C, Nikayin S, Misak CJ, Flood PD, Kiedrowski K, Alhazzani W. Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2018 Sep;46(9):e825-e873. doi: 10.1097/CCM.0000000000003299. PMID 30113379
- [Background] Riker RR, Picard JT, Fraser GL. Prospective evaluation of the Sedation-Agitation Scale for adult critically ill patients. Crit Care Med. 1999 Jul;27(7):1325-9. doi: 10.1097/00003246-199907000-00022. PMID 10446827
- [Background] Sessler CN, Gosnell MS, Grap MJ, Brophy GM, O'Neal PV, Keane KA, Tesoro EP, Elswick RK. The Richmond Agitation-Sedation Scale: validity and reliability in adult intensive care unit patients. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1338-44. doi: 10.1164/rccm.2107138. PMID 12421743
- [Background] Balzer F, Weiss B, Kumpf O, Treskatsch S, Spies C, Wernecke KD, Krannich A, Kastrup M. Early deep sedation is associated with decreased in-hospital and two-year follow-up survival. Crit Care. 2015 Apr 28;19(1):197. doi: 10.1186/s13054-015-0929-2. PMID 25928417
- [Background] Shehabi Y, Bellomo R, Reade MC, Bailey M, Bass F, Howe B, McArthur C, Seppelt IM, Webb S, Weisbrodt L; Sedation Practice in Intensive Care Evaluation (SPICE) Study Investigators; ANZICS Clinical Trials Group. Early intensive care sedation predicts long-term mortality in ventilated critically ill patients. Am J Respir Crit Care Med. 2012 Oct 15;186(8):724-31. doi: 10.1164/rccm.201203-0522OC. Epub 2012 Aug 2. PMID 22859526
- [Background] Kollef MH, Levy NT, Ahrens TS, Schaiff R, Prentice D, Sherman G. The use of continuous i.v. sedation is associated with prolongation of mechanical ventilation. Chest. 1998 Aug;114(2):541-8. doi: 10.1378/chest.114.2.541. PMID 9726743
- [Background] Kress JP, Pohlman AS, O'Connor MF, Hall JB. Daily interruption of sedative infusions in critically ill patients undergoing mechanical ventilation. N Engl J Med. 2000 May 18;342(20):1471-7. doi: 10.1056/NEJM200005183422002. PMID 10816184
- [Background] Shehabi Y, Bellomo R, Reade MC, Bailey M, Bass F, Howe B, McArthur C, Murray L, Seppelt IM, Webb S, Weisbrodt L; Sedation Practice in Intensive Care Evaluation Study Investigators; Australian and New Zealand Intensive Care Society Clinical Trials Group. Early goal-directed sedation versus standard sedation in mechanically ventilated critically ill patients: a pilot study*. Crit Care Med. 2013 Aug;41(8):1983-91. doi: 10.1097/CCM.0b013e31828a437d. PMID 23863230
- [Background] Rampil IJ. A primer for EEG signal processing in anesthesia. Anesthesiology. 1998 Oct;89(4):980-1002. doi: 10.1097/00000542-199810000-00023. No abstract available. PMID 9778016
- [Background] Hemmerling TM, Charabati S, Bracco D. Unusual case of low bispectral index values due to electrocardiographic interferences. Br J Anaesth. 2008 Dec;101(6):877-8. doi: 10.1093/bja/aen289. No abstract available. PMID 19004916
- [Background] Vretzakis G, Dragoumanis C, Ferdi H, Papagiannopoulou P. Influence of an external pacemaker on bispectral index. Eur J Anaesthesiol. 2005 Jan;22(1):70-2. doi: 10.1017/s0265021505230144. No abstract available. PMID 15816579
- [Background] Schuller PJ, Newell S, Strickland PA, Barry JJ. Response of bispectral index to neuromuscular block in awake volunteers. Br J Anaesth. 2015 Jul;115 Suppl 1:i95-i103. doi: 10.1093/bja/aev072. PMID 26174308
- [Background] Vereecke HE, Struys MM, Mortier EP. A comparison of bispectral index and ARX-derived auditory evoked potential index in measuring the clinical interaction between ketamine and propofol anaesthesia. Anaesthesia. 2003 Oct;58(10):957-61. doi: 10.1046/j.1365-2044.2003.03403.x. PMID 12969037
- [Background] Messner M, Beese U, Romstock J, Dinkel M, Tschaikowsky K. The bispectral index declines during neuromuscular block in fully awake persons. Anesth Analg. 2003 Aug;97(2):488-491. doi: 10.1213/01.ANE.0000072741.78244.C0. PMID 12873942
- [Background] Gurudatt C. Sedation in Intensive Care Unit patients: Assessment and awareness. Indian J Anaesth. 2011 Nov;55(6):553-5. doi: 10.4103/0019-5049.90607. No abstract available. PMID 22223896
- [Background] Vender JS, Szokol JW, Murphy GS, Nitsun M. Sedation, analgesia, and neuromuscular blockade in sepsis: an evidence-based review. Crit Care Med. 2004 Nov;32(11 Suppl):S554-61. doi: 10.1097/01.ccm.0000145907.86298.12. PMID 15542964
- [Background] Shetty RM, Bellini A, Wijayatilake DS, Hamilton MA, Jain R, Karanth S, Namachivayam A. BIS monitoring versus clinical assessment for sedation in mechanically ventilated adults in the intensive care unit and its impact on clinical outcomes and resource utilization. Cochrane Database Syst Rev. 2018 Feb 21;2(2):CD011240. doi: 10.1002/14651858.CD011240.pub2. PMID 29464690
- [Background] Boncompte G, Sun H, Elgueta MF, Benavides J, Carrasco M, Morales MI, Calderon N, Contreras V, Westover MB, Cortinez LI, Akeju O, Pedemonte JC. Intraoperative electroencephalographic marker of preoperative frailty: A prospective cohort study. J Clin Anesth. 2023 Jun;86:111069. doi: 10.1016/j.jclinane.2023.111069. Epub 2023 Feb 2. PMID 36738630
- [Background] Biggs D, Boncompte G, Pedemonte JC, Fuentes C, Cortinez LI. The effect of age on electroencephalogram measures of anesthesia hypnosis: A comparison of BIS, Alpha Power, Lempel-Ziv complexity and permutation entropy during propofol induction. Front Aging Neurosci. 2022 Aug 11;14:910886. doi: 10.3389/fnagi.2022.910886. eCollection 2022. PMID 36034131
- [Background] Ali HH, Utting JE, Gray C. Stimulus frequency in the detection of neuromuscular block in humans. 1970. Br J Anaesth. 1998 Apr;80(4):530-41; discussion 528-9. doi: 10.1093/bja/80.4.530. No abstract available. PMID 9640166
- [Background] Thilen SR, Weigel WA, Todd MM, Dutton RP, Lien CA, Grant SA, Szokol JW, Eriksson LI, Yaster M, Grant MD, Agarkar M, Marbella AM, Blanck JF, Domino KB. 2023 American Society of Anesthesiologists Practice Guidelines for Monitoring and Antagonism of Neuromuscular Blockade: A Report by the American Society of Anesthesiologists Task Force on Neuromuscular Blockade. Anesthesiology. 2023 Jan 1;138(1):13-41. doi: 10.1097/ALN.0000000000004379. PMID 36520073
- [Background] Simonetti M, Ceron C, Galiano A, Lake ET, Aiken LH. Hospital work environment, nurse staffing and missed care in Chile: A cross-sectional observational study. J Clin Nurs. 2022 Sep;31(17-18):2518-2529. doi: 10.1111/jocn.16068. Epub 2021 Oct 4. PMID 34723415
- [Background] Rasulo FA, Hopkins P, Lobo FA, Pandin P, Matta B, Carozzi C, Romagnoli S, Absalom A, Badenes R, Bleck T, Caricato A, Claassen J, Denault A, Honorato C, Motta S, Meyfroidt G, Radtke FM, Ricci Z, Robba C, Taccone FS, Vespa P, Nardiello I, Lamperti M. Processed Electroencephalogram-Based Monitoring to Guide Sedation in Critically Ill Adult Patients: Recommendations from an International Expert Panel-Based Consensus. Neurocrit Care. 2023 Apr;38(2):296-311. doi: 10.1007/s12028-022-01565-5. Epub 2022 Jul 27. PMID 35896766
- [Background] Purdon PL, Pavone KJ, Akeju O, Smith AC, Sampson AL, Lee J, Zhou DW, Solt K, Brown EN. The Ageing Brain: Age-dependent changes in the electroencephalogram during propofol and sevoflurane general anaesthesia. Br J Anaesth. 2015 Jul;115 Suppl 1(Suppl 1):i46-i57. doi: 10.1093/bja/aev213. PMID 26174300
- [Background] Purdon PL, Sampson A, Pavone KJ, Brown EN. Clinical Electroencephalography for Anesthesiologists: Part I: Background and Basic Signatures. Anesthesiology. 2015 Oct;123(4):937-60. doi: 10.1097/ALN.0000000000000841. PMID 26275092
- [Background] Hight DF, Kaiser HA, Sleigh JW, Avidan MS. Continuing professional development module : An updated introduction to electroencephalogram-based brain monitoring during intended general anesthesia. Can J Anaesth. 2020 Dec;67(12):1858-1878. doi: 10.1007/s12630-020-01820-3. Epub 2020 Nov 15. PMID 33190217
- [Background] Tse AHW, Ling L, Lee A, Joynt GM. Altered Pharmacokinetics in Prolonged Infusions of Sedatives and Analgesics Among Adult Critically Ill Patients: A Systematic Review. Clin Ther. 2018 Sep;40(9):1598-1615.e2. doi: 10.1016/j.clinthera.2018.07.021. Epub 2018 Aug 31. PMID 30173953
- [Background] Hanidziar D, Bittner EA. Sedation of Mechanically Ventilated COVID-19 Patients: Challenges and Special Considerations. Anesth Analg. 2020 Jul;131(1):e40-e41. doi: 10.1213/ANE.0000000000004887. No abstract available. PMID 32392023
- [Background] Hanidziar D, Westover MB. Monitoring of sedation in mechanically ventilated patients using remote technology. Curr Opin Crit Care. 2022 Jun 1;28(3):360-366. doi: 10.1097/MCC.0000000000000940. PMID 35653256
- [Background] Nagaraj SB, Biswal S, Boyle EJ, Zhou DW, McClain LM, Bajwa EK, Quraishi SA, Akeju O, Barbieri R, Purdon PL, Westover MB. Patient-Specific Classification of ICU Sedation Levels From Heart Rate Variability. Crit Care Med. 2017 Jul;45(7):e683-e690. doi: 10.1097/CCM.0000000000002364. PMID 28441231
- [Background] Raj R, Ussavarungsi K, Nugent K. Accelerometer-based devices can be used to monitor sedation/agitation in the intensive care unit. J Crit Care. 2014 Oct;29(5):748-52. doi: 10.1016/j.jcrc.2014.05.014. Epub 2014 May 28. PMID 24973100
- [Background] Wennervirta JE, Sarkela MOK, Kaila MM, Pettila V. Responsiveness Index versus the RASS-Based Method for Adjusting Sedation in Critically Ill Patients. Crit Care Res Pract. 2021 Oct 7;2021:6621555. doi: 10.1155/2021/6621555. eCollection 2021. PMID 34659830
- [Background] Zheng WL, Sun H, Akeju O, Westover MB. Adaptive Sedation Monitoring From EEG in ICU Patients With Online Learning. IEEE Trans Biomed Eng. 2020 Jun;67(6):1696-1706. doi: 10.1109/TBME.2019.2943062. Epub 2019 Sep 23. PMID 31545708
- [Background] Sun H, Kimchi E, Akeju O, Nagaraj SB, McClain LM, Zhou DW, Boyle E, Zheng WL, Ge W, Westover MB. Automated tracking of level of consciousness and delirium in critical illness using deep learning. NPJ Digit Med. 2019 Sep 9;2:89. doi: 10.1038/s41746-019-0167-0. eCollection 2019. PMID 31508499
- [Background] Tonna JE, Dalton A, Presson AP, Zhang C, Colantuoni E, Lander K, Howard S, Beynon J, Kamdar BB. The Effect of a Quality Improvement Intervention on Sleep and Delirium in Critically Ill Patients in a Surgical ICU. Chest. 2021 Sep;160(3):899-908. doi: 10.1016/j.chest.2021.03.030. Epub 2021 Mar 24. PMID 33773988
- [Background] Fahy BG, Chau DF. The Technology of Processed Electroencephalogram Monitoring Devices for Assessment of Depth of Anesthesia. Anesth Analg. 2018 Jan;126(1):111-117. doi: 10.1213/ANE.0000000000002331. PMID 28786839
- [Background] Weber F, Seidl M, Bein T. Impact of the AEP-Monitor/2-derived composite auditory-evoked potential index on propofol consumption and emergence times during total intravenous anaesthesia with propofol and remifentanil in children. Acta Anaesthesiol Scand. 2005 Mar;49(3):277-83. doi: 10.1111/j.1399-6576.2005.00626.x. PMID 15752388
- [Background] Cortinez LI, Delfino AE, Fuentes R, Munoz HR. Performance of the cerebral state index during increasing levels of propofol anesthesia: a comparison with the bispectral index. Anesth Analg. 2007 Mar;104(3):605-10. doi: 10.1213/01.ane.0000255152.96354.17. PMID 17312217
- [Background] Viertio-Oja H, Maja V, Sarkela M, Talja P, Tenkanen N, Tolvanen-Laakso H, Paloheimo M, Vakkuri A, Yli-Hankala A, Merilainen P. Description of the Entropy algorithm as applied in the Datex-Ohmeda S/5 Entropy Module. Acta Anaesthesiol Scand. 2004 Feb;48(2):154-61. doi: 10.1111/j.0001-5172.2004.00322.x. No abstract available. PMID 14995936
- [Background] Revuelta M, Paniagua P, Campos JM, Fernandez JA, Martinez A, Jospin M, Litvan H. Validation of the index of consciousness during sevoflurane and remifentanil anaesthesia: a comparison with the bispectral index and the cerebral state index. Br J Anaesth. 2008 Nov;101(5):653-8. doi: 10.1093/bja/aen245. Epub 2008 Aug 23. PMID 18723856
- [Background] Kreuer S, Wilhelm W. The Narcotrend monitor. Best Pract Res Clin Anaesthesiol. 2006 Mar;20(1):111-9. doi: 10.1016/j.bpa.2005.08.010. PMID 16634418
- [Background] Zikov T, Bibian S, Dumont GA, Huzmezan M, Ries CR. Quantifying cortical activity during general anesthesia using wavelet analysis. IEEE Trans Biomed Eng. 2006 Apr;53(4):617-32. doi: 10.1109/TBME.2006.870255. PMID 16602568
- [Background] Drover D, Ortega HR. Patient state index. Best Pract Res Clin Anaesthesiol. 2006 Mar;20(1):121-8. doi: 10.1016/j.bpa.2005.07.008. PMID 16634419
- [Background] Willmann K, Springman S, Rusy D, Daily E. A preliminary evaluation of a new derived EEG index monitor in anesthetized patients. J Clin Monit Comput. 2002 Aug;17(6):345-50. doi: 10.1023/a:1024266026091. PMID 12885178
- [Background] Jensen EW, Valencia JF, Lopez A, Anglada T, Agusti M, Ramos Y, Serra R, Jospin M, Pineda P, Gambus P. Monitoring hypnotic effect and nociception with two EEG-derived indices, qCON and qNOX, during general anaesthesia. Acta Anaesthesiol Scand. 2014 Sep;58(8):933-41. doi: 10.1111/aas.12359. Epub 2014 Jul 4. PMID 24995461
- [Background] Fritz BA, Kalarickal PL, Maybrier HR, Muench MR, Dearth D, Chen Y, Escallier KE, Ben Abdallah A, Lin N, Avidan MS. Intraoperative Electroencephalogram Suppression Predicts Postoperative Delirium. Anesth Analg. 2016 Jan;122(1):234-42. doi: 10.1213/ANE.0000000000000989. PMID 26418126
- [Background] Soehle M, Dittmann A, Ellerkmann RK, Baumgarten G, Putensen C, Guenther U. Intraoperative burst suppression is associated with postoperative delirium following cardiac surgery: a prospective, observational study. BMC Anesthesiol. 2015 Apr 28;15:61. doi: 10.1186/s12871-015-0051-7. PMID 25928189
- [Background] Pedemonte JC, Plummer GS, Chamadia S, Locascio JJ, Hahm E, Ethridge B, Gitlin J, Ibala R, Mekonnen J, Colon KM, Westover MB, D'Alessandro DA, Tolis G, Houle T, Shelton KT, Qu J, Akeju O. Electroencephalogram Burst-suppression during Cardiopulmonary Bypass in Elderly Patients Mediates Postoperative Delirium. Anesthesiology. 2020 Aug;133(2):280-292. doi: 10.1097/ALN.0000000000003328. PMID 32349072
- [Background] Zhang XS, Roy RJ, Jensen EW. EEG complexity as a measure of depth of anesthesia for patients. IEEE Trans Biomed Eng. 2001 Dec;48(12):1424-33. doi: 10.1109/10.966601. PMID 11759923
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. Ann Intern Med. 2007 Oct 16;147(8):573-7. doi: 10.7326/0003-4819-147-8-200710160-00010. PMID 17938396
- [Background] Ely EW, Margolin R, Francis J, May L, Truman B, Dittus R, Speroff T, Gautam S, Bernard GR, Inouye SK. Evaluation of delirium in critically ill patients: validation of the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). Crit Care Med. 2001 Jul;29(7):1370-9. doi: 10.1097/00003246-200107000-00012. PMID 11445689
- [Background] Donoghue T, Haller M, Peterson EJ, Varma P, Sebastian P, Gao R, Noto T, Lara AH, Wallis JD, Knight RT, Shestyuk A, Voytek B. Parameterizing neural power spectra into periodic and aperiodic components. Nat Neurosci. 2020 Dec;23(12):1655-1665. doi: 10.1038/s41593-020-00744-x. Epub 2020 Nov 23. PMID 33230329
- [Background] Wiest C, Torrecillos F, Pogosyan A, Bange M, Muthuraman M, Groppa S, Hulse N, Hasegawa H, Ashkan K, Baig F, Morgante F, Pereira EA, Mallet N, Magill PJ, Brown P, Sharott A, Tan H. The aperiodic exponent of subthalamic field potentials reflects excitation/inhibition balance in Parkinsonism. Elife. 2023 Feb 22;12:e82467. doi: 10.7554/eLife.82467. PMID 36810199
- [Background] Stam CJ, Nolte G, Daffertshofer A. Phase lag index: assessment of functional connectivity from multi channel EEG and MEG with diminished bias from common sources. Hum Brain Mapp. 2007 Nov;28(11):1178-93. doi: 10.1002/hbm.20346. PMID 17266107
- [Background] Brown EN, Lydic R, Schiff ND. General anesthesia, sleep, and coma. N Engl J Med. 2010 Dec 30;363(27):2638-50. doi: 10.1056/NEJMra0808281. No abstract available. PMID 21190458
- [Background] Kaiser HA, Hirschi T, Sleigh C, Reineke D, Hartwich V, Stucki M, Rummel C, Sleigh J, Hight D. Comorbidity-dependent changes in alpha and broadband electroencephalogram power during general anaesthesia for cardiac surgery. Br J Anaesth. 2020 Oct;125(4):456-465. doi: 10.1016/j.bja.2020.06.054. Epub 2020 Jul 31. PMID 32747077
- [Background] Massimini M, Ferrarelli F, Huber R, Esser SK, Singh H, Tononi G. Breakdown of cortical effective connectivity during sleep. Science. 2005 Sep 30;309(5744):2228-32. doi: 10.1126/science.1117256. PMID 16195466
- [Background] Ferrarelli F, Massimini M, Sarasso S, Casali A, Riedner BA, Angelini G, Tononi G, Pearce RA. Breakdown in cortical effective connectivity during midazolam-induced loss of consciousness. Proc Natl Acad Sci U S A. 2010 Feb 9;107(6):2681-6. doi: 10.1073/pnas.0913008107. Epub 2010 Jan 25. PMID 20133802
- [Background] Sarasso S, Rosanova M, Casali AG, Casarotto S, Fecchio M, Boly M, Gosseries O, Tononi G, Laureys S, Massimini M. Quantifying cortical EEG responses to TMS in (un)consciousness. Clin EEG Neurosci. 2014 Jan;45(1):40-9. doi: 10.1177/1550059413513723. Epub 2014 Jan 8. PMID 24403317
- [Background] Jospin M, Caminal P, Jensen EW, Litvan H, Vallverdu M, Struys MM, Vereecke HE, Kaplan DT. Detrended fluctuation analysis of EEG as a measure of depth of anesthesia. IEEE Trans Biomed Eng. 2007 May;54(5):840-6. doi: 10.1109/TBME.2007.893453. PMID 17518280
- [Background] Cortinez LI, Anderson BJ, Penna A, Olivares L, Munoz HR, Holford NH, Struys MM, Sepulveda P. Influence of obesity on propofol pharmacokinetics: derivation of a pharmacokinetic model. Br J Anaesth. 2010 Oct;105(4):448-56. doi: 10.1093/bja/aeq195. Epub 2010 Aug 14. PMID 20710020
- [Background] Bjelland TW, Klepstad P, Haugen BO, Nilsen T, Dale O. Effects of hypothermia on the disposition of morphine, midazolam, fentanyl, and propofol in intensive care unit patients. Drug Metab Dispos. 2013 Jan;41(1):214-23. doi: 10.1124/dmd.112.045567. Epub 2012 Oct 31. PMID 23115086
- [Background] Saeed M, Villarroel M, Reisner AT, Clifford G, Lehman LW, Moody G, Heldt T, Kyaw TH, Moody B, Mark RG. Multiparameter Intelligent Monitoring in Intensive Care II: a public-access intensive care unit database. Crit Care Med. 2011 May;39(5):952-60. doi: 10.1097/CCM.0b013e31820a92c6. PMID 21283005
- [Background] Hyun DG, Ahn JH, Gil HY, Nam CM, Yun C, Lim CM. Longitudinal trajectories of sedation level and clinical outcomes in patients who are mechanically ventilated based on a group-based trajectory model: a prospective, multicentre, longitudinal and observational study in Korea. BMJ Open. 2023 Jun 27;13(6):e072628. doi: 10.1136/bmjopen-2023-072628. PMID 37369420
- [Background] Kang J, Cho YS, Lee M, Yun S, Jeong YJ, Won YH, Hong J, Kim S. Effects of nonpharmacological interventions on sleep improvement and delirium prevention in critically ill patients: A systematic review and meta-analysis. Aust Crit Care. 2023 Jul;36(4):640-649. doi: 10.1016/j.aucc.2022.04.006. Epub 2022 Jun 17. PMID 35718628
- [Background] Fiest KM, Soo A, Hee Lee C, Niven DJ, Ely EW, Doig CJ, Stelfox HT. Long-Term Outcomes in ICU Patients with Delirium: A Population-based Cohort Study. Am J Respir Crit Care Med. 2021 Aug 15;204(4):412-420. doi: 10.1164/rccm.202002-0320OC. PMID 33823122
- [Background] Salluh JI, Wang H, Schneider EB, Nagaraja N, Yenokyan G, Damluji A, Serafim RB, Stevens RD. Outcome of delirium in critically ill patients: systematic review and meta-analysis. BMJ. 2015 Jun 3;350:h2538. doi: 10.1136/bmj.h2538. PMID 26041151
- [Background] Stollings JL, Kotfis K, Chanques G, Pun BT, Pandharipande PP, Ely EW. Delirium in critical illness: clinical manifestations, outcomes, and management. Intensive Care Med. 2021 Oct;47(10):1089-1103. doi: 10.1007/s00134-021-06503-1. Epub 2021 Aug 16. PMID 34401939